CLINICAL TRIAL: NCT01705522
Title: Multimodal Approach in IBD Patients
Acronym: MAID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinical Hospital Colentina (Other)
Responsible Party: Principal Investigator, dr. Theodor Alexandru Voiosu, Gastroenterology resident, Teaching Assistant, Clinical Hospital Colentina
Other Study IDs: COL-GASTRO-3
Record Dates: First submitted 2012-10-10; First posted 2012-10-12 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Ulcerative Colitis; Crohn's Disease; Nonalcoholic Fatty Liver Disease (NAFLD); Vitamin D Deficiency
Keywords: IBD; ulcerative colitis; Crohn's disease; NAFLD; biomarkers; vitamin D
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Non-alcoholic Fatty Liver Disease; Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and fecal samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IBD patients: patients with ulcerative colitis or crohn's disease, in remission

SUMMARY:
The investigators intend to assess the role of several biomarkers in the prediction of relapse in IBD. Clinical, laboratory and endoscopic data will be gathered and a predictive score will be derived in order to assess the relapse risk at 1 year.

DETAILED DESCRIPTION:
Patients with a confirmed diagnosis of IBD will be prospectively assessed on a yearly basis in order to assess relapse risk factors.

Disease activity will be assessed using the Mayo score for UC patients and CDAI for Crohn's disease and endoscopic activity will be assessed using the Mayo endoscopic subscore for UC patients and the Simple Endoscopic Score for Crohn's Disease for CD patients.

Serum and fecal biomarkers will be obtainted at each study visit (C-reactive protein, fecal calprotectin).

Data about current and past medication for IBD will also be gathered.

ELIGIBILITY:
Inclusion Criteria:

* ulcerative colitis or Crohn's disease
* age over 18
* clinical remission
* signed informed consent

Exclusion Criteria:

* pregnant women
* refusal to sign informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients with IBD over 18 years of age, currently in clinical remission
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-10; Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Clinical relapse | 1 year
  clinical relapse as assessed by conventional scores for activity in IBD - Mayo or CDAI
Prevalence of NAFLD | 1 year
  to assess the prevalence of nonalcoholic liver disease in IBD patients
prevalence of vitamin D deficiency | 1 year
  to assess vitamin D deficiency and osteopenia among IBD patients

CONTACTS AND LOCATIONS:
Overall Officials: Theodor Voiosu, Md, Principal Investigator — Clinical Hospital Colentina
Locations (1):
- Colentina Clinical Hospital, Bucharest, Romania

REFERENCES:
- [Background] Dionne S, Hiscott J, D'Agata I, Duhaime A, Seidman EG. Quantitative PCR analysis of TNF-alpha and IL-1 beta mRNA levels in pediatric IBD mucosal biopsies. Dig Dis Sci. 1997 Jul;42(7):1557-66. doi: 10.1023/a:1018895500721. PMID 9246063
- [Derived] Voiosu T, Bengus A, Dinu R, Voiosu AM, Balanescu P, Baicus C, Diculescu M, Voiosu R, Mateescu B. Rapid fecal calprotectin level assessment and the SIBDQ score can accurately detect active mucosal inflammation in IBD patients in clinical remission: a prospective study. J Gastrointestin Liver Dis. 2014 Sep;23(3):273-8. doi: 10.15403/jgld.2014.1121.233.thv. PMID 25267955